CLINICAL TRIAL: NCT01037972
Title: Influence of Whole Body Vibration Compared to Conventional Physiotherapy in Patients With Gonarthrosis
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Gregor Stein, Dr. med, University of Cologne
Other Study IDs: Galileo; 2009-017617-29 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
Keywords: Galileo; Whole body vibration; Osteoarthritis; Knee; Physiotherapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Whole body vibration
  Interventions: Behavioral: Whole body vibration
- Conventional physiotherapy
  Interventions: Behavioral: Conventional physiotherapy

INTERVENTIONS:
Behavioral: Conventional physiotherapy — 3 times weekly 30 minutes of conventional physiotherapy to strengthen muscular strength and balance in the lower extremity.
  Other Names: Galileo
  Groups: Conventional physiotherapy
Behavioral: Whole body vibration — 3 times weekly 30 minutes of exercises on a whole body vibration device to strengthen muscular strength and improve muscular balance in the lower extremity.
  Other Names: Galileo Whole body vibration
  Groups: Whole body vibration

SUMMARY:
40 patients with osteoarthritis of the knee will be randomly assigned to conventional physiotherapy on the one and whole body vibration exercises on the other hand. The duration of the training will be 6 weeks, three times a week.

The outcome will be measured by WOMAC and SF-12 scores relating to pain and quality of life. The second outcome criteria will be a motion analysis and balance testing before and after the training.

The follow-up is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 30-80 years old
* WOMAC 30-70 mm (VAS)
* Gonarthrosis (Kellgren/Lawrence) II-III

Exclusion Criteria:

* WOMAC >70 mm (VAS)
* Endoprosthesis in lower extremity
* BMI >40 kg/m2

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis of the knee.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 6 weeks after inclusion

SECONDARY OUTCOMES:
Motion analysis | 6 weeks after inclusion
Pain reduction | 12 weeks after inclusion
Pain reduction | 26 weeks after inclusion
Motion analysis | 12 weeks after inclusion
Motion analysis | 26 weeks after inclusion
Quality of life | 6 weeks after inclusion
Quality of life | 12 weeks after inclusion
Quality of life | 26 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Zarghooni, MD, Principal Investigator — University of Cologne; Gregor Stein, MD, Study Director — University of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Stein G, Knoell P, Faymonville C, Kaulhausen T, Siewe J, Otto C, Eysel P, Zarghooni K. Whole body vibration compared to conventional physiotherapy in patients with gonarthrosis: a protocol for a randomized, controlled study. BMC Musculoskelet Disord. 2010 Jun 21;11:128. doi: 10.1186/1471-2474-11-128. PMID 20565956
- See also: University Hospital of Cologne — http://www.uk-koeln.de